CLINICAL TRIAL: NCT03296956
Title: A Dietary Supplement for Mood Symptoms in Early Postpartum: A Double Blind Randomized Placebo Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Jeff Meyer, Program Head, Neurochemical Imaging for Mood Disorders, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 083/2015
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Postpartum Blues; Healthy
Keywords: Postpartum; Dietary Supplement; Mood Symptoms

STUDY DESIGN:
Intervention Model Description: one arm receives Motherwell and one arm receives placebo; randomized double blind The supplement is expected to prevent depressed mood induction during postpartum blues whereas the placebo is not. The effect of depressed mood induction is strong during postpartum blues in 75% to 95% of mothers (who do not take Motherwell). The supplement is the intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: all are blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Day-5 postpartum - Active dietary supplement (Active Comparator): Healthy women on day-5 postpartum. This group is recruited during pregnancy but the main study day, involving the dietary supplement consumption is being done after delivery and during postpartum.
  Intervention: Full dose dietary supplement Motherwell
  Interventions: Dietary Supplement: Motherwell
- Day-5 postpartum - Placebo (Placebo Comparator): Healthy women on day-5 postpartum. This group is recruited during pregnancy but the main study day, involving the dietary supplement consumption is being done after delivery and during postpartum.
  Intervention: Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Motherwell — The interventions involves a dietary supplement called Motherwell, at current stage, to reduce the intensity of sadness in day-5 postpartum women.
  Arms: Day-5 postpartum - Active dietary supplement
Other: Placebo — Matching placebo for appearance, taste
  Arms: Day-5 postpartum - Placebo

SUMMARY:
The purpose of this study is to determine whether a dietary supplement (DS) is effective in protecting against sad mood in postpartum as compared to placebo.

DETAILED DESCRIPTION:
This double blind placebo controlled randomized trial will evaluate the effect of administration of a dietary supplement (DS) on the intensity of postpartum blues. It is expected that the administration will result in less sadness in day-5 postpartum women after negative mood induction in those receiving the dietary supplement compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45
* BMI 19 to 40 (kg/m2)
* Resting pulse between 45 and 100 bpm
* Systolic blood pressure between 91 and 139 mmHg (inclusive)
* Diastolic blood pressure between 51 and 90 mmHg (inclusive)
* Orthostatic blood pressure change <20 mmHg (based on the difference between supine and standing (1 minute) systolic blood pressure)

Exclusion Criteria:

* The subject has been diagnosed with any axis 1 and 2 disorders based on Structured Clinical Interview (SCID) for the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5) interview within the past 10 years.
* Subjects who have been smoking cigarettes in the past 5 years (to reduce variability in mood attributable to cigarette withdrawal and monoamine oxidase A (MAO-A)).
* Intolerance to any of the components of the intervention.
* If in the principal investigator's judgement the obstetric or neonatal complications were so severe that would cause change in the results of the study, such as infant death, the subject will be excluded.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) | Assessment will be done on day-5 postpartum. On the assessment day, the VAS will be administered before and after sad mood induction and compared]
  VAS uses a 10-cm scale for participants to indicate the extent to which each of them feel happy or sad. The change in VAS before versus after sad mood induction is the change score in VAS. The change score on the day with active dietary supplement is compare to the change score of the subjects who have received placebo

SECONDARY OUTCOMES:
Change in Profile of Mood States (POMS) Scores | Assessment will be done on day-5 postpartum. On the assessment day, the POMS will be administered before and after sad mood induction and compared]
  The POMS contains 65 adjectives rated by participants on a 5-point scale. Six factors are derived that include tension, depression, anger, fatigue, vigor and confusion

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H Meyer, MD,PhD,FRCPC, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiciton and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dowlati Y, Ravindran AV, Segal ZV, Stewart DE, Steiner M, Meyer JH. Selective dietary supplementation in early postpartum is associated with high resilience against depressed mood. Proc Natl Acad Sci U S A. 2017 Mar 28;114(13):3509-3514. doi: 10.1073/pnas.1611965114. Epub 2017 Mar 13. PMID 28289215
- [Background] Dowlati Y, Ravindran AV, Maheux M, Steiner M, Stewart DE, Meyer JH. No effect of oral L-tryptophan or alpha-lactalbumin on total tryptophan levels in breast milk. Eur Neuropsychopharmacol. 2015 Jun;25(6):779-87. doi: 10.1016/j.euroneuro.2015.03.005. Epub 2015 Mar 18. PMID 25823693
- [Background] Dowlati Y, Ravindran AV, Maheux M, Steiner M, Stewart DE, Meyer JH. No effect of oral tyrosine on total tyrosine levels in breast milk: implications for dietary supplementation in early postpartum. Arch Womens Ment Health. 2014 Dec;17(6):541-8. doi: 10.1007/s00737-014-0441-8. PMID 25015680
- [Background] Sacher J, Wilson AA, Houle S, Rusjan P, Hassan S, Bloomfield PM, Stewart DE, Meyer JH. Elevated brain monoamine oxidase A binding in the early postpartum period. Arch Gen Psychiatry. 2010 May;67(5):468-74. doi: 10.1001/archgenpsychiatry.2010.32. PMID 20439828
- [Background] Meyer JH, Wilson AA, Sagrati S, Miler L, Rusjan P, Bloomfield PM, Clark M, Sacher J, Voineskos AN, Houle S. Brain monoamine oxidase A binding in major depressive disorder: relationship to selective serotonin reuptake inhibitor treatment, recovery, and recurrence. Arch Gen Psychiatry. 2009 Dec;66(12):1304-12. doi: 10.1001/archgenpsychiatry.2009.156. PMID 19996035
- [Background] Meyer JH, Ginovart N, Boovariwala A, Sagrati S, Hussey D, Garcia A, Young T, Praschak-Rieder N, Wilson AA, Houle S. Elevated monoamine oxidase a levels in the brain: an explanation for the monoamine imbalance of major depression. Arch Gen Psychiatry. 2006 Nov;63(11):1209-16. doi: 10.1001/archpsyc.63.11.1209. PMID 17088501
- [Derived] Meyer JH, Wang Z, Santhirakumar A, Dowlati Y, Docteur N, Shoaib A, Purnava J, Wang Y, Wang W, Chen S, Husain MI, de Silva Wijeyeratne R, Reeyaz H, Baena-Tan C, Koshimori Y, Nasser Z, Sit V. Dietary supplement for mood symptoms in early postpartum: a double-blind randomized placebo controlled trial. EClinicalMedicine. 2024 Apr 10;71:102593. doi: 10.1016/j.eclinm.2024.102593. eCollection 2024 May. PMID 38813444